CLINICAL TRIAL: NCT04166695
Title: Clinical Performance of Long-span All-ceramic or Metal-ceramic Fixed Partial Dentures on Implants and/or Natural Teeth
Brief Title: Clinical Performance of Long-span Fixed Partial Dentures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Dr. Wolfgang Bömicke, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-682/2019
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monolithic / facially veneered zirconia (Experimental): Participants receive one monolithic / facially veneered zirconia fixed partial denture.
  Interventions: Device: Monolithic / facially veneered zirconia fixed partial denture
- Completely veneered CoCr (Other): Control group. Participants receive one completely veneered metal ceramic fixed partial denture.
  Interventions: Device: Completely veneered CoCr fixed partial denture

INTERVENTIONS:
Device: Monolithic / facially veneered zirconia fixed partial denture — Participant receives one monolithic / facially veneered zirconia fixed partial denture retained by either teeth, implants or teeth and implants for the replacement of two neighbouring posterior teeth.
  Arms: Monolithic / facially veneered zirconia
Device: Completely veneered CoCr fixed partial denture — Participant receives one completely veneered CoCr fixed partial denture retained by either teeth, implants or teeth and implants for the replacement of two neighbouring posterior teeth.
  Arms: Completely veneered CoCr

SUMMARY:
Tooth-coloured fixed restorations are becoming increasingly popular with patients and dentists. If high-strength all-ceramics such as zirconia are used as the restoration material, a maximum of two adjacent missing teeth can be replaced with the aid of fixed partial dentures (FPDs). For the replacement of a missing anterior or posterior tooth by FPDs, a very good clinical performance similar to that of metal-based, ceramic-veneered restorations can be expected. However, evidence-based statements on the clinical performance of long-span all-ceramic FPDs are difficult because there are only very few studies on this topic, which are also inhomogeneous with regard to the study conditions. Randomized studies to compare monolithic (consisting only of the high-strength framework material) or partially veneered (weaker veneering ceramics in esthetically relevant tooth areas) all-ceramic and classic (completely veneered) metal-ceramic FPDs are lacking. The aim of the current explorative, prospective, randomized, two-arm clinical interventional study is therefore to compare the clinical performance of long-span FPDs (≥ 4 Pontics) made of monolithic / facially veneered zirconium dioxide with a gold standard (completely veneered cobalt chromium (CoCr)-based FPDs). Forty patients will be recruited. Once all inclusion criteria have been established, including the signed informed consent of the patients informed of the content, effort, advantages and disadvantages of the study, patients are assigned to the two study groups by stratified block randomization (main strata: tooth-supported / (tooth-)implant-supported). After placement of the restorations, follow-up examinations are performed after 1 week (baseline) and after half a year, one year, two years and three years. In addition to the main target criterion (veneering defects), further complications (related to FPDs or supporting tissues / structures) and parameters of oral health are recorded. Depending on the distribution and structure of the data, parametric and non-parametric statistics are used. Group differences with respect to the main target criterion ceramic defects are to be investigated by log-rank and chi-square tests. The significance level is set at α < 0.05. Since this is an explorative study, all p-values are descriptive.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years old.
* The patient has unrestricted legal capacity.
* The patient has two posterior teeth (premolars and / or molars) that are to be replaced next to each other.
* The patient is reliable and willing to take part in follow-up examinations regularly and over the entire study period (three years).
* The information about the study has been understood by the patient and the signed declaration of consent has been received.

Exclusion Criteria:

* Pregnancy and lactation
* Local and / or systemic acute and / or chronic (also in the past) general medical diseases and conditions that contradict participation in the study and / or expose the patient to a higher risk in the case of participation in the study.
* Severe bruxism diagnosed by a portable electrocardiomyography device (BruxOff) (> 4 bruxism episodes / night)
* Reduced clinical crown height (< 5 mm before tooth preparation)
* Limited periodontal health:

  * probing depths > 4 mm or = 4 mm and bleeding on probing,
  * Furcation involvement > I (first band of the periodontometer after Naber disappears completely)
  * Degree of loosening of the abutment teeth > Grade I (> 1 mm horizontal mobility)
* Untreated endodontic problems of abutment teeth
* Lack of antagonistic support from fixed dentures or natural teeth
* Known allergies or intolerances to the materials used in the study
* Lack of oral hygiene
* Lack of compliance
* Planned change of residence
* Rejection of randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time-dependent ceramic defect rate | 3 years
  The time to the occurrence of a ceramic defect is used as the main target criterion. Ceramic defects are identified in a structured clinical examination after cleaning and drying of the restoration surface and with the aid of magnifying glasses.

SECONDARY OUTCOMES:
Restoration survival | 3 years
  Time-dependent survival rate
Abutment-tooth survival | 3 years
  Time-dependent survival rate of abutment teeth
Implant survival | 3 years
  Time-dependent survival rate of implants
Restoration success | 3 years
  Time-dependent complication-free survival rate of restorations
Abutment-tooth success | 3 years
  Time-dependent complication-free survival rate of abutment teeth
Implant success | 3 years
  Time-dependent complication-free survival rate of implants
Risk-factor analysis | 3 years
  Identification of influencing factors (risk factors such as sex, the position of the fixed partial denture in the upper or lower jaw, a tooth or implant-supported design, and the activity of the masticatory muscles) for the occurrence of complications.
Gingival / mucosal, periodontal / periimplant health of the abutment teeth / implants | 3 years
  The gingival / mucosal inflammation is evaluated categorically (0 - 3) on the basis of the gingival index (GI) according to Loe and Silness. Periodontal / periimplant health is assessed by measuring the pocket depth around teeth and implants using a millimeter-scaled periodontal probe and by simultaneously measuring the incidence of bleeding on probing (BOP) and suppuration.
Plaque accumulation | 3 years
  The accumulation of dental / peri-implant plaque is determined categorically (0 - 3) on the basis of the Plaque Index (PI) according to Silness and Loe.
Patients' satisfaction with restoration esthetics | 3 years
  Satisfaction with the esthetics of the restorations is assessed by the patient on a 6-point visual analogue scale.
Wear on the restoration and the natural opposing dentition | 3 years
  Quantification of the clinical wear (vertical height loss and volume loss) that has occurred on the restorations and antagonistic material using 3D superimposed diagnostic models

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Bömicke, PD Dr. MSc., Principal Investigator — Department of Prosthodontics, University Hospital Heidelberg, University of Heidelberg
Locations (1):
- Department of Prosthodontics, University Hospital Heidelberg, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany